CLINICAL TRIAL: NCT00289796
Title: Assess the Feasibility of an Investigational Vaccination Regimen, Compared to a 3-dose Primary Vaccination With GSK Biologicals' Infanrix Hexa™ (DTPa-HBV-IPV/Hib Vaccine) Following Hepatitis B Vaccination at Birth. Primary Vaccination is Followed in the 2nd Year of Life by a Booster Dose of Infanrix-hexa
Brief Title: Assess Feasibility of an Acellular Pertussis Vaccine (Pa) Given Soon After Birth, Followed by 3-dose Primary Vaccination With the DTPa-HBV-IPV/Hib Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 210602-002; 105752 (Other: GSK)
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Infanrix hexa Group (Active Comparator): Subjects received a dose of hepatitis B vaccine at birth followed by immunization with 3 doses of Infanrix hexa™ (2, 4 and 6 months of age) and one booster dose of Infanrix hexa™ between 12 and 23 months of age. All vaccines were administered by deep intramuscular injection into the left anterolateral thigh.
  Interventions: Biological: DTPa-HBV-IPV/Hib

INTERVENTIONS:
Biological: DTPa-HBV-IPV/Hib — GSK Biologicals' combined diphtheria, tetanus, acellular pertussis, hepatitis B, inactivated poliovirus and Haemophilus influenzae type b conjugate vaccine

SUMMARY:
This study will assess immunogenicity, safety and reactogenicity of primary and booster vaccination.

DETAILED DESCRIPTION:
"There will be two groups in this study:

* one group will receive a birth dose of Pa vaccine and 3 doses of DTPa-HBV-IPV/Hib vaccine as primary vaccination and a dose of DTPa-HBV-IPV/Hib vaccine as booster vaccination
* the control group will receive a birth dose of hepatitis B vaccine and 3 doses of DTPa-HBV-IPV/Hib vaccine as primary vaccination and a dose of DTPa-HBV-IPV/Hib vaccine as booster vaccination".

ELIGIBILITY:
Inclusion criteria For the primary vaccination phase

* Healthy newborn male or female infant 2 to 5 days old at the time of the first vaccination & written informed consent taken from the parents/guardians of the subject
* Born at term (gestational age 37-42 weeks) after an uncomplicated pregnancy
* Birth weight >= 2.5 kg and 5 minute Apgar >= 7
* Mother seronegative for Hepatitis B surface antigen (HBsAg) For the booster vaccination phase
* A healthy male or female between, and including, 12 and 23 months of age at the time of booster vaccination who has completed the primary vaccination course in the primary vaccination phase with written informed consent obtained from the parent or guardian of the subject

Exclusion criteria For the primary vaccination phase

* Mother known or suspected to be seropositive for HIV (testing not required for inclusion)
* Planned use of any investigational or non-registered product (drug or vaccine) other than the study vaccines during the study
* Planned administration of immuno-suppressants or other immune-modifying drugs, administration of immunoglobulins and/or any blood products since birth or planned administration during the study.
* Administration of immunoglobulins and/or any blood products to the mother during pregnancy
* Neonatal jaundice requiring parenteral treatment (light therapy for physiological jaundice is allowed)
* At risk of pneumococcal disease or planning to receive Prevenar™ during the study period
* Administration or planned administration of BCG vaccination during the study period
* Acute disease at the time of vaccination. For the booster vaccination phase
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the booster dose, or planned use during the booster phase.
* Evidence of previous diphtheria, tetanus, pertussis, polio, hepatitis B and/or Hib booster vaccination since the study conclusion visit of the primary vaccination phase.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* Administration/ planned administration of a vaccine not foreseen by the study protocol, administration/ planned administration of immunoglobulins and/or any blood products during the period starting 30 days before the administration of the booster dose and ending 30 days after the booster dose.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the booster vaccine dose."

Ages: 2 Days to 5 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2004-07; Primary Completion 2006-04 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of seropositive subjects for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 0
  A seropositive subject was defined a subject with antibody concentrations ≥ 5 EL.U/mL.
Number of seropositive subjects for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 3
  A seropositive subject was defined a subject with antibody concentrations ≥ 5 EL.U/mL.
Number of seropositive subjects for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 5
  A seropositive subject was defined a subject with antibody concentrations ≥ 5 EL.U/mL.
Number of seropositive subjects for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 7
  A seropositive subject was defined a subject with antibody concentrations ≥ 5 EL.U/mL.
Antibody concentrations for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 0
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off of ≥ 5 EL.U/mL.
Antibody concentrations for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 3
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off of ≥ 5 EL.U/mL.
Antibody concentrations for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 5
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off of ≥ 5 EL.U/mL.
Antibody concentrations for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 7
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off of ≥ 5 EL.U/mL.
Number of seropositive subjects for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 1 Post-Booster
  A seropositive subject was defined a subject with antibody concentrations ≥ 5 EL.U/mL.
Antibody concentrations for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 1 Post-Booster
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seropositivity cut-off of ≥ 5 EL.U/mL.
Modified vaccine response for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 7
  Modified vaccine response was defined as: For initially seronegative subjects, antibody concentration 5 EL.U/mL at one month after the third dose of Infanrix hexa™. For initially seropositive subjects: antibody concentration at one month post vaccination 0.25 fold the pre-vaccination antibody concentration.
Modified vaccine response for anti-pertussis toxoids (PT), anti-filamentous hemagglutinin (FHA) and anti-pertactin (PRN) antibodies | At Month 1 Post-Booster
  Modified vaccine response was defined as: For initially seronegative subjects, antibody concentration 5 EL.U/mL at one month after the third dose of Infanrix hexa™. For initially seropositive subjects: antibody concentration at one month post vaccination 0.25 fold the pre-vaccination antibody concentration.
Number of seroprotected subjects for anti-Hepatitis B surface antigen (anti-HBs) antibodies | At Month 7
  A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/mL.
Number of seroprotected subjects for anti-Hepatitis B surface antigen (anti-HBs) antibodies | At pre-booster vaccination (Month 0 BST)
  A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/mL.
Number of seroprotected subjects for anti-Hepatitis B surface antigen (anti-HBs) antibodies | At Month 1 post-booster vaccination
  A seroprotected subject was defined as a subject with anti-HBs antibody concentrations ≥ 10 mIU/mL.
Antibody concentrations for anti-Hepatitis B surface antigen (anti-HBs) antibodies | At Month 7
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 10 mIU/mL.
Antibody concentrations for anti-Hepatitis B surface antigen (anti-HBs) antibodies | At pre-booster vaccination (Month 0 BST)
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 10 mIU/mL.
Antibody concentrations for anti-Hepatitis B surface antigen (anti-HBs) antibodies | At Month 1 post-booster vaccination
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 10 mIU/mL.
Number of seroprotected subjects for anti-diphtheria (anti-D) and anti-tetanus (anti-T) antibodies | At Month 7
  A seroprotected subject was defined as a subject with anti-D and anti-T antibody concentrations ≥ 0.1 IU/mL.
Number of seroprotected subjects for anti-diphtheria (anti-D) and anti-tetanus (anti-T) antibodies | At pre-booster vaccination (Month 0 BST)
  A seroprotected subject was defined as a subject with anti-D and anti-T antibody concentrations ≥ 0.1 IU/mL.
Number of seroprotected subjects for anti-diphtheria (anti-D) and anti-tetanus (anti-T) antibodies | At Month 1 post-booster vaccination
  A seroprotected subject was defined as a subject with anti-D and anti-T antibody concentrations ≥ 0.1 IU/mL.
Antibody concentrations for anti-diphtheria (anti-D) and anti-tetanus (anti-T) antibodies | At Month 7
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 0.1 IU/mL.
Antibody concentrations for anti-diphtheria (anti-D) and anti-tetanus (anti-T) antibodies | At pre-booster vaccination (Month 0 BST)
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 0.1 IU/mL.
Antibody concentrations for anti-diphtheria (anti-D) and anti-tetanus (anti-T) antibodies | At Month 1 post-booster vaccination
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 0.1 IU/mL.
Number of seroprotected subjects for anti-polyribosyl ribitol phosphate (anti-PRP) | At Month 7
  A seroprotected subject was defined as a subject with anti-D and anti-T antibody concentrations ≥ 0.15 g/mL.
Number of seroprotected subjects for anti-polyribosyl ribitol phosphate (anti-PRP) | At pre-booster vaccination (Month 0 BST)
  A seroprotected subject was defined as a subject with anti-D and anti-T antibody concentrations ≥ 0.15 g/mL.
Number of seroprotected subjects for anti-polyribosyl ribitol phosphate (anti-PRP) | At Month 1 post-booster vaccination
  A seroprotected subject was defined as a subject with anti-D and anti-T antibody concentrations ≥ 0.15 g/mL.
Antibody concentrations for anti-polyribosyl ribitol phosphate (anti-PRP) | At Month 7
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 0.15 g/mL.
Antibody concentrations for anti-polyribosyl ribitol phosphate (anti-PRP) | At pre-booster vaccination (Month 0 BST)
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 0.15 g/mL.
Antibody concentrations for anti-polyribosyl ribitol phosphate (anti-PRP) | At Month 1 post-booster vaccination
  Concentrations were expressed as geometric mean concentrations (GMCs) for the seroprotection cut-off of ≥ 0.15 g/mL.
Number of subjects with solicited general symptoms | During the 8-day (Day 0-Day 7) follow-up period after the any dose and booster vaccination
  The solicited local symptoms assessed were Drowsiness, Temperature (Fever), Irritability and Loss of appetite. Temperature = Fever ≥ 38.0 °C. Grade 3 drowsiness = drowsiness that prevented normal activity; Grade 3 irritability = crying that could not be comforted/prevented normal activity; Grade 3 loss of appetite = not eating at all; Grade 3 Temperature = > 39.5 °C. Related = symptoms considered by the investigator to have a causal relationship to vaccination.
Number of subjects with unsolicited adverse events (AES) | Occurring within Day 0-30 following primary and booster vaccination
  An AE was defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Knuf M, Schmitt HJ, Wolter J, Schuerman L, Jacquet JM, Kieninger D, Siegrist CA, Zepp F. Neonatal vaccination with an acellular pertussis vaccine accelerates the acquisition of pertussis antibodies in infants. J Pediatr. 2008 May;152(5):655-60, 660.e1. doi: 10.1016/j.jpeds.2007.09.034. Epub 2007 Nov 19. PMID 18410769
- [Background] Knuf M, Schmitt HJ, Jacquet JM, Collard A, Kieninger D, Meyer CU, Siegrist CA, Zepp F. Booster vaccination after neonatal priming with acellular pertussis vaccine. J Pediatr. 2010 Apr;156(4):675-8. doi: 10.1016/j.jpeds.2009.12.019. PMID 20303444
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 210602-002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 210602-002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 210602-002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 210602-002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 210602-002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 210602-002 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register